CLINICAL TRIAL: NCT06093750
Title: Correlation Between State-Trait-Anxiety-Inventory and Heart Rate Variability: An Observational Cohort and Pilot Study
Brief Title: Correlation Between State-Trait-Anxiety-Inventory and Heart Rate Variability
Status: Completed | Type: Observational
Sponsor: Ludwig Boltzmann Institute for Traumatology - The research center in cooperation with AUVA (Other Government)
Collaborators: UKH Salzburg (Unknown); University of Ulm (Other); Institute for Salutology (Unknown)
Responsible Party: Sponsor
Other Study IDs: Version 1.2
Record Dates: First submitted 2023-10-04; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Preoperative Vegetative Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to investigate whether there is a correlation between the vegetative stress evaluated by the State-Trait-Anxiety-Inventory (STAI-Test) and the measurement of heart rate variability (HRV). A subgroup analysis will also be performed to determine whether premedication contributes to a lower STAI score and/or heart rate variability. The primary outcome will be the parameter of frequency-based analysis Low Frequency (LF) and High Frequency (HF), and the STAI score. Secondary outcomes are the parameters Low Frequency/High Frequency-ratio (LF/HF-ratio), Standard deviation of normal-to-normal (NN) intervals (SDNN), Root Mean Square of successive differences" (RMSSD) and mean heart rate, age, gender, if they are smokers and if they work in shifts.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 65 years
* Elective surgery with a low risk of bleeding
* American Society of Anesthesiologists (ASA) classification 1-2
* metabolic equivalent of task (MET) > 4

Exclusion Criteria:

* Pre-existing cardiac conditions such as heart failure, arterial hypertension,
* diabetes
* any central nervous system diseases
* cardiac pacemaker
* renal and hepatic insufficiency
* regional or peridural anesthesia
* Pregnancy, lactation
* Drugs that directly influence the autonomic nervous system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects are recruited after the anesthesia interview with the anesthesiologist.
  anesthesiologist. Subjects with elective surgery associated with a low risk of bleeding will be included. This includes procedures such as knee arthroplasties, cruciate ligamentoplasties, or metal removals.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
State and Trait Anxiety Inventory (STAI-score) | First questionnaire is given 40 minutes before transfer to the holding area and the second questionnaire postoperative in the recovery ward directly before transfer back to ward
  STAI: State-Trait-Anxiety-Inventory-Score This test consists of 40 items and assesses the current state of anxiety in relation to the current situation in which the patient is to the current situation in which the patient finds herself (State Anxiety) and the general anxiety state existing state of anxiety, which represents a part of her personality (Trait Anxiety). A score of 20-80 could be achieved, with higher scores correlating with correlated with higher anxiety levels. Accordingly, scores of 20-39, 40-59, and 60-80 would indicate low, moderate, and high anxiety.
The measurement method of heart rate variability (especially the parameter of the frequency domain Low Frequency and High Frequency | One measurement (3-6 hours), start of measurement together with the first STAI questionnaire (40 min before transfer to the holding area), end of measurement after the second STAI questionnaire is done.
  Low frequency power (LF):
  Power density spectrum in the frequency range from 0.04-0.15 Hz
  High frequency power (HF):
  Power density spectrum in the frequency range from 0.15 to 0.40 Hz

SECONDARY OUTCOMES:
Heart rate variability ("Standard deviation of normal-to-normal (NN) intervals" (SDNN) and "Root Mean Square of successive differences" (RMSSD) of the time domain and "LF/HF-ratio" from the frequency domain) as well as mean heart rate | HRV-parameters and mean heart rate were obtained in the same time frame as outcome 2.
  Standard deviation of NN-intervals (SDNN):
  intervals in the measuring range; NN-intervals refer to the intervals between normal R-peaks in an electrocardiogram
  Root Mean Square of successive differences (RMSSD)
  Low Frequency/High Frequency-ratio (LF/HF ratio):
  Quotient of the spectrum in LF and the spectrum in HF, No clear assignment, Ratio or Coefficient or Ratio between LF-and HF Band power
Age, gender, if they are smokers and if they work in shifts | Outcomes will be collected following the routine anaesthesia interview with the anaesthesiologist as part of the recruitment process.
  Age: 18-65
  Gender: male, female
  smoker: no, (never; nonsmoker > 1 year), yes (< 5/d; 6-15/d; >15/d)
  working in shifts: yes, no

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Fritsch, PD. Dr., Principal Investigator — Ludwig Boltzmann Institute for Traumatology - The research center in cooperation with AUVA
Locations (1):
- Allgemeine Unfallversicherungsanstalt, Salzburg, Austria